CLINICAL TRIAL: NCT02766673
Title: Safety and Efficacy of Aerosolized Albuterol in Mechanically Ventilated Infants With Bronchopulmonary Dysplasia (BDP)
Brief Title: Aerosolized Albuterol Use in Severe BPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-012264
Record Dates: First submitted 2016-05-09; First posted 2016-05-10 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Severe Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full Dose Albuterol Sulfate (Active Comparator): 2.5mg of Albuterol Sulfate will be administered via nebulizer and mechanical ventilator
  Interventions: Drug: Albuterol Sulfate
- Half Dose Albuterol Sulfate (Active Comparator): 1.25mg of Albuterol Sulfate will be administered via nebulizer and mechanical ventilator
  Interventions: Drug: Albuterol Sulfate
- Sterile Saline (Placebo Comparator): 3ml of 0.9% sterile saline will be administered via nebulizer and mechanical ventilator
  Interventions: Drug: Sterile Saline

INTERVENTIONS:
Drug: Albuterol Sulfate — Subjects will receive a dose of study medication every 4 hours for 24 total hours
  Other Names: Salbutamol
  Arms: Full Dose Albuterol Sulfate; Half Dose Albuterol Sulfate
Drug: Sterile Saline — Subjects will receive a dose of study medication every 4 hours for 24 total hours
  Other Names: Placebo
  Arms: Sterile Saline

SUMMARY:
Currently several dose schedules of Albuterol are administered via nebulization to infants in the neonatal and infant intensive care unit (N/IICU). As Albuterol is not FDA approved for this population (under 2 years) there is no standard recommended dose. Aerosolized Albuterol is one of the most widely used therapies that are utilized for infants with chronic lung disease. The common practice in the N/IICU is weight base dosing of all medications. This contradicts the aerosol science recommendations, which advise not to titrate doses by weight as the patient naturally self-regulates their dose according to the change in minute ventilation with age. In addition, the wide use of aerosolized Albuterol in the infant with Bronchopulmonary Dysplasia (BPD) has little current evidence of efficacy in this disease. Understanding the appropriate dose for effective treatment as well as the indication for use in the BPD population would provide the clinician with useful guidelines.

The investigators propose to analyze the safety and efficacy of aerosolized albuterol in infants with BPD comparing the recommended dose per aerosolization literature with the common dosing practices at The Children's Hospital of Philadelphia (CHOP) as well as placebo.

DETAILED DESCRIPTION:
This is a randomized, blinded cross-over study of infants with a diagnosis of Severe BPD that are mechanically ventilated. Participants will receive 3 sets of treatment (2.5mg Albuterol, 1.25mg Albuterol, 3ml normal saline placebo), in random order. Each treatment will be administered every 4 hours for 24 hours. After a 6 hour washout phase, the next group of interventions will be applied. Following another wash-out phase, the final group of intervention will be applied. Pulmonary mechanics from the ventilator (e.g. airway compliance, airway resistance, tidal volume, peak inspiratory pressure, Forced Expiratory Flow at 75% of forced vital capacity, etc.) and the patient short term response to therapy (heart rate, blood pressure, heart rhythm) will be assessed for the duration of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Infants greater than or equal to 36 weeks corrected gestational age to one year of age
2. Diagnosis of BPD in accordance with The Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) definition
3. May have a current order for short acting bronchodilator, not required
4. May have congenital anomalies unless one or more of the exclusion criteria are met, not required
5. Receiving conventional mechanical ventilation via an artificial airway (endotracheal tube or tracheostomy) via Draeger V500 Ventilator
6. Parental/guardian permission (informed consent)

Exclusion Criteria:

1. Airway leak greater than 10%
2. Unilateral lung disease
3. Current order for inhaled anticholinergic (i.e. ipratropium bromide)
4. Active pulmonary or systemic infection
5. Scheduled order for other medication that cause bronchodilation (i.e. atrovent, magnesium sulfate, ketamine, etc.)

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Dysart, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original study sample size called for 25 subjects. The block randomization scheme of 6 treatment sequences within 1 randomization block. Therefore we recruited 24 patients to complete 4 randomization block. the 25th patient would have started a new randomization block and make one treatment sequence more common that the others.
Groups:
- Treatment Sequence A: Treatment group 1: Placebo (0.9% sterile saline) every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 2: 1.25mg Albuterol every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 3: 2.5 mg Albuterol every 4 hours for 24 hours
- Treatment Sequence B: Treatment group 1: Placebo (0.9% sterile saline) every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 2: 2.5mg Albuterol every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 3: 1.25mg Albuterol every 4 hours for 24 hours
- Treatment Sequence C: Treatment Group 1: 1.25 mg Albuterol every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 2: Placebo (0.9% sterile saline) every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 3: 2.5mg albuterol every 4 hours for 24 hours
- Treatment Sequence D: Treatment Group 1: 1.25 mg Albuterol every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 2: 2.5mg albuterol every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 3: Placebo (0.9% sterile saline) every 4 hours for 24 hours
- Treatment Sequence E: Treatment group 1: 2.5mg albuterol every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 2: Placebo (0.9% sterile saline) every 4 hours for 24 hours
  6 hour washout phase
  Treatment Group 3: 1.25 mg Albuterol every 4 hours for 24 hours
- Treatment Sequence F: Treatment group 1: 2.5mg albuterol every 4 hours for 24 hours
  6 hour washout phase
  Treatment Group 2: 1.25 mg Albuterol every 4 hours for 24 hours
  6 hour washout phase
  Treatment group 3: Placebo (0.9% sterile saline) every 4 hours for 24 hours
Period: Overall Study
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C | Treatment Sequence D | Treatment Sequence E | Treatment Sequence F
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4 | 4 | 3
Not Completed | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This was a crossover study therefore all patients were scheduled to receive all 3 treatment groups. Enrollment demographics will be the same for all groups.
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: days] | 170.4 (49.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 4
  More than one race | 0
  Unknown or Not Reported | 11
Weight [Mean (Standard Deviation); unit: kg] | 4.7 (1.5)
Birth Gestational Age [Mean (Standard Deviation); unit: weeks] | 25 (1.9)
Birth Weight [Median (Standard Deviation); unit: g] | 611 (12)
Corrected Gestational Age [Mean (Standard Deviation); unit: Weeks] | 49 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Expiratory Flow Between Pre and Post-medication Dosing
Description: Expiratory flow at 75% of vital capacity (EF75) will be measured before beginning each treatment and again 15-30 min after each treatment phase. Therefore there will be 6 pairs (12) of EF values to determine the change in EF for each treatment. this measure is done by measuring the expiratory flow at 75% of exhalation on as measure on the flow volume loop of the ventilator. a single mechanical breath is chosen and the flow volume loop is frozen on the ventilator screen. the clinician can then scroll to measure total tidal volume for the breath, then multiple this volume by 0.25 (to ascertain the volume that the time point of 75% of exhalation), then scroll along the expiratory side of the flow volume loop until the calculated volume is reached and then the flow at that time point is recorded.
Time Frame: every 4 hours in each treatment group, up to 24 hours
Population: Each subject had the potential for 6 paired observations (12 measures) per treatment group (comparison of measure before and after each dose of the study drug). 2 subjects did not complete all 3 treatment groups. Some measurements were missed leaving less than the total potential number of observations.
Measure: Mean (Standard Deviation); unit: L/min
Units Other Than Participants: EF 75% Observatrions
Arm/Group | Full Dose Albuterol Sulfate | Half Dose Albuterol Sulfate | Sterile Saline
Number analyzed (Participants) | 23 | 23 | 23
Number analyzed (EF 75% Observatrions) | 129 | 141 | 134
L/min | 0.38 (2.3) | 0.70 (2.4) | 0.45 (2.5)

2. Secondary Outcome: Percent Change in Heart Rate (Beats/Min) Between Pre and Post-medication Dosing
Description: Heart rate will be measured before beginning each treatment and again 15-30 min after the conclusion of each treatment phase (4 hours). Therefore there will be 6 pairs of heart rates (12 measures), to determine the change in HR for each treatment group.
Time Frame: every 4 hours in each treatment group, up to 24 hours
Population: There was a potential for up to 6 paired observations (12 measures) per treatment group. 2 patients did not complete all 3 treatment groups resulting is lower number of observations for the potential total.
Measure: Mean (Standard Deviation); unit: % change
Units Other Than Participants: Heart Rate measurements beats/min
Arm/Group | Full Dose Albuterol Sulfate | Half Dose Albuterol Sulfate | Sterile Saline
Number analyzed (Participants) | 23 | 23 | 23
Number analyzed (Heart Rate measurements beats/min) | 132 | 144 | 138
% change | 0.074 (0.129) | 0.031 (0.120) | 0.009 (0.084)

ADVERSE EVENTS:
Time Frame: Adverse events were continuously monitored for and were attributed to a given treatment group from the time that the first treatment was given through the washout phase following the given treatment group. Albuterol has an effect range for 4-6 hours so any adverse events from the medication. Time frame of monitoring for adverse events ended 6 hours after the final medication dose was administered.
Groups:
- Full Dose Albuterol: 2.5mg of Albuterol Sulfate will be administered via nebulizer and mechanical ventilator
  Albuterol Sulfate: Subjects will receive a dose of study medication every 4 hours for 24 total hours
- Half Dose Albuterol: 1.25mg of Albuterol Sulfate will be administered via nebulizer and mechanical ventilator
  Albuterol Sulfate: Subjects will receive a dose of study medication every 4 hours for 24 total hours
Arm/Group | Full Dose Albuterol | Half Dose Albuterol | Sterile Saline
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT02766673/Prot_SAP_000.pdf